CLINICAL TRIAL: NCT04769934
Title: Impact of Implant Insertion Torque on Peri-implant Bone Level.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Irena Sailer, Prof. Dr. Irena Sailer, Head of the Division, University of Geneva, Switzerland
Other Study IDs: 2018-00666
Record Dates: First submitted 2021-02-17; First posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Implant Complication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Penguin RFA — to evaluate the peri-implant bone level changes (marginal bone level) around the implant platform.

SUMMARY:
Observational study with one single arm. The purpose of this study was to evaluate the impact of the insertion torque and of the implant stability on the marginal bone level changes for dental implants placed into healed ridges.

DETAILED DESCRIPTION:
The primary outcome would be to evaluate the peri-implant bone level changes (marginal bone level) around the implant platform.

The secondary outcomes would be:

* To evaluate the Implant Stability Quotient (ISQ) changes according to the measurements performed with the instrument Penguin RFA
* To evaluate the implant and prosthetic failure rate as well as the implant and prosthetic complication rates
* The patient satisfaction related to the implant treatment

ELIGIBILITY:
Inclusion Criteria:

* All partially edentulous patients requiring simple Implant placement,
* being at least 18-year-old and able to sign an informed consent,
* The patients that will be enrolled must have a bone quantity that allows the placement of regular implants according to the radiographic evaluations (pre-operative radiographic examination).

Exclusion Criteria:

* Heavy smokers (more than 10 cigarettes/day).
* Immunosuppressed or immunocompromised patients
* Uncontrolled diabetes
* Active periodontal disease
* Patients with a full mouth marginal bleeding score higher than 20%
* Addiction to alcohol or drugs
* Psychiatric problems
* Severe caries, periapical lesions, acute infection (abscess)
* Immediate post-extractive implants (at least 2 months after extraction have to elapse)
* Patients unable to commit to 3-year follow-up.
* Patients treated or under treatment with intravenous amino- bisphosphonates.
* Patients participating to other studies, if the present protocol could not be fully adhered to.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: partially edentulous patients
Sampling Method: Non-Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
radiographic marginal bone level changes around the implant platform | 3 years
  the changes (in mm) of the marginal bone level around the implant platform

SECONDARY OUTCOMES:
Implant Stability Quotient (ISQ) changes | 3 years
  the measurements will be performed with the instrument Penguin RFA

OTHER OUTCOMES:
implant failure rate | 3 years
  % of implant failure
patient satisfaction related to the implant treatment | 3 years
  degree of satisfaction on factors such as function, comfort and esthetics through questionnaires
prosthetic failure rate | 3 years
  % of prosthetic failure
implant complications rate | 3 years
  % of implant complications
prosthetic complications rate | 3 years
  % of prosthetic complications

CONTACTS AND LOCATIONS:
Overall Officials: Irena Sailer, Prof. Dr., Principal Investigator — University of Geneva
Locations (1):
- University of Geneva, Geneva, Switzerland